CLINICAL TRIAL: NCT06894173
Title: EvoLution of Neoadjuvant TreatMent in 'Triple-negative' or 'HER-2-positive' Breast Cancer Diagnosed in the EaRly Phase: Retrospective Multicentre Study on the Therapeutic Approach Most Commonly Adopted in the Italian Oncology Centres
Brief Title: EvoLution of Neoadjuvant TreatMent in 'Triple-negative' or 'HER-2-positive' Breast Cancer Diagnosed in the EaRly Phase
Acronym: GIM28-ELMER
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4946
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to describe the percentage of patients with HER2-positive and Triple Negative tumour underwent neoadjuvant treatment in clinical practice during the past 5 years out of total number of patients who underwent neoadjuvant treatment, regardless molecular subtypes. Secondary objectives The secondary objectives which are limited to molecular subtypes of study interest, HER2-positive and Triple Negative tumours, are follow reported:

* To perform a descriptive analysis on neoadjuvant treatment choice according to molecular subtype and initial staging;
* To perform a descriptive analysis on clinical and tumour pathological characteristics according to molecular subtypes and initial staging;
* To perform radiological response descriptive analysis achieved with neoadjuvant therapy according to treatment and instrumental examination type (for example: breast MRI, breast ultrasound or mammography);
* To perform a descriptive analysis of surgical procedures for both, the breast and the axilla, according to radiological tumour response, initial staging and molecular subtypes;
* To perform a descriptive analysis on therapies performed in adjuvant setting according to neoadjuvant treatment type, initial staging and molecular subtypes;
* To describe and to analyse the eligibility criteria evolution in neoadjuvant treatment setting during the last 5 years;
* To perform a descriptive analysis on pathological complete response (cPR) according to neoadjuvant treatment, molecular subtypes and initial staging;
* To evaluate disease-free survival (DFS) according to pCR and molecular subtypes;
* To evaluate overall survival (OS) according to pCR and molecular subtypes.

ELIGIBILITY:
Inclusion Criteria:

* For primary endpoint assessment we calculated the percentage of HER2 positive and Triple Negative patients who underwent neoadjuvant treatment in the past 5 years in each site. For this aim all patients with early breast cancer diagnosis who underwent neoadjuvant treatment during the study time, ranging from 01/01/2016 to 01/01/2021, will be included if they had:
* Histological diagnosis of infiltrating breast cancer performed by breast and/or axillary nodes biopsy;
* Age ≥ 18 years at the time of disease onset;
* Absence of secondary lesions, i.e. initial disease stage I, II or III;
* Known status of ER, PgR, HER-2 and Ki67.

Exclusion Criteria:

* Documented distant disease at onset diagnosis or within 3 months from breast surgery;
* Prior neoadjuvant hormonal treatment exposure;
* Prior diagnosis of primary breast cancer or second primitive tumour starting from different organ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for this retrospective, non-interventional study, must have been exposed to neoadjuvant chemotherapy with or without target therapies in the 5-year period from 01/01/2016 to 01/01/2021
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-03 (Actual); Primary Completion 2025-12-03 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with HER2-positive and Triple Negative tumour among early breast cancer who underwent neoadjuvant treatment | 5 years
  The primary endpoint will express as the ratio between the total number of patients with HER2-positive and TN tumour who underwent neoadjuvant treatment out of total number of patients who had early breast cancer diagnosis and who underwent neoadjuvant treatment during the entire study time, regardless molecular subtype. The primary endpoint will be calculated according molecular subtypes, as follow specified: 'Luminal a and b', 'Triple Negative', 'HER-2 enriched' and 'HER-2 luminal'. The molecular subtypes will be identified and classified according to the 2018 American Society of Clinical Oncology and College of American Pathologists (ASCO-CAP) definition.

SECONDARY OUTCOMES:
The frequency of different treatments used in neoadjuvant setting according to initial staging and molecular subtypes; | 5 years
  HER-2 positive and Triple Negative patients subtypes.
The frequency of different clinical and pathological tumour characteristics according to initial staging and molecular subtypes; | 5 years
  HER-2 positive and Triple Negative patients
The frequency of complete radiological response according to neoadjuvant treatment, instrumental examination (breast MRI, breast ultrasound or mammography) used in clinical practice and molecular subtypes; | 5 years
  HER-2 positive and Triple Negative patients
The frequency of different surgical procedures for both, the breast and the axilla, according to radiological response, initial staging and molecular subtypes; | 5 years
  HER-2 positive and Triple Negative patients
The frequency of different treatments adopted in adjuvant setting according to neoadjuvant treatment type, initial staging and molecular subtypes. | 5 years
  HER-2 positive and Triple Negative patients
The frequency of pathologic complete response (pCR) according to molecular subtypes and neoadjuvant treatment; | 5 years
  HER-2 positive and Triple Negative patients
Descriptive analysis of the correlation between complete radiologic response and pCR according to molecular subtypes and neoadjuvant treatment. | 5 years
  HER-2 positive and Triple Negative patients
Descriptive analysis of the correlation between pCR and DFS according to the different molecular subtypes. | 5 years
  HER-2 positive and Triple Negative patients. DFS will be calculated as time interval from the date of first neoadjuvant cycle to the date of onset disease recurrence at local, contralateral or at distance level. For patients without recurrence at the time of DFS analysis, the second date will be censored at the time of last control.
Correlation analysis between pCR and OS according to the different molecular subtypes. | 5 years
  HER-2 positive and Triple Negative patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Fabi, Principal Investigator — Fondazione Policlinico Universitario A.Gemelli IRCCS, UOC Senologia; Antonella Palazzo, Principal Investigator — Fondazione Policlinico Universitario A.Gemelli IRCCS, UOC Oncologia Medica
Locations (29):
- Italy (29):
  - IRCCS - Centro di Riferimento Oncologico (C.R.O.) di Aviano, Aviano, PN
  - AOU Ospedali Riuniti Torrette di Ancona, Ancona
  - A.O.R.N. "San Giuseppe Moscati", Avellino
  - Presidio di Brindisi Di Summa - Perrino, Brindisi
  - Humanitas Istituto Clinico Catanese, Catania
  - Azienda Ospedaliera Universitaria "San Martino" - Istituto Nazionale per la Ricerca sul Cancro, Genova
  - ASST - Azienda Ospedaliera Carlo Poma di Mantova, Mantova
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST S.r.l., Meldola
  - Istituto Europeo di Oncologia, Milan
  - ASST - Ospedale Sacco, Milan
  - Azienda Ospedaliera Universitaria - P.O. di Modena, Modena
  - Azienda Ospedaliera "A. Cardarelli", Napoli
  - Istituto Nazionale Tumori di Napoli - IRCCS Istituto Pascale, Napoli
  - Universita' degli Studi di Napoli Federico II, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliera Regionale San Carlo, Potenza
  - Nuovo Ospedale di Prato - S. Stefano, Prato
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - AOU Policlinico Umberto I, Roma
  - Ospedale Sandro Pertini - ASL Roma 2, Roma
  - Fondazione Policlinico A. Gemelli, IRCCS, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Arcispedale di Santo Spirito in Sassia - Nuovo Regina Margherita, Roma
  - Azienda Socio Sanitaria Territoriale ( ASST ) della Valtellina e Alto Lario Presidio di Sondalo, Sondalo
  - A.O.U. Città della salute e della scienza - Presidio Molinette, Torino
  - APSS - Ospedale Santa Chiara di Trento, Trento
  - Ospedale di Belcolle - Viterbo, Viterbo

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.